CLINICAL TRIAL: NCT03726879
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Clinical Trial To Evaluate the Efficacy and Safety Of Atezolizumab or Placebo in Combination With Neoadjuvant Doxorubicin + Cyclophosphamide Followed By Paclitaxel + Trastuzumab + Pertuzumab In Early Her2-Positive Breast Cancer
Brief Title: A Study To Evaluate the Efficacy and Safety Of Atezolizumab or Placebo in Combination With Neoadjuvant Doxorubicin + Cyclophosphamide Followed By Paclitaxel + Trastuzumab + Pertuzumab In Early Her2-Positive Breast Cancer
Acronym: IMpassion050
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BO40747
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Results first posted 2022-03-25 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — atezolizumab; Doxorubicin; Cyclophosphamide; Paclitaxel; Trastuzumab; pertuzumab; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atezolizumab +ddAC-PacHP (Experimental): Participants will receive atezolizumab (atezo) 840 mg IV Q2W for 4 cycles during neoadjuvant phase with ddAC (doxorubicin 60 mg/m2 & cyclophosphamide 600 mg/m2 IV), followed by atezo 1200 mg IV Q3W for 4 cycles with paclitaxel 80 mg/m2 IV weekly for 12 continuous weeks, trastuzumab 6 mg/kg IV (with initial 8mg/kg IV loading dose) Q3W for 4 cycles, & pertuzumab 420 mg IV (with initial 840-mg IV loading dose) Q3W for 4 cycles. During adjuvant phase, participants will continue to receive following study treatments Q3W to complete up to 1 year HER2-target therapy inclusive of therapy given both in neoadjuvant and adjuvant setting: atezo 1200 mg IV Q3W, trastuzumab 6 mg/kg IV (with initial 8-mg/kg IV loading dose) Q3W, & pertuzumab 420 mg IV (with initial 840-mg IV loading dose) Q3W. Participants who do not achieve pCR have option of receiving blinded atezo+trastuzumab emtansine post surgery for 14 cycles. In response to USM DIL dated 3 Feb 2021 treatment with atezo must be discontinued.
  Interventions: Drug: Atezolizumab; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Trastuzumab Emtansine
- Placebo + ddAC-PacHP (Placebo Comparator): Participants will receive placebo 840 mg IV Q2W for 4 cycles during neoadjuvant phase with ddAC (doxorubicin 60 mg/m2 & cyclophosphamide 600 mg/m2 IV), followed by placebo 1200 mg IV Q3W for 4 cycles with paclitaxel 80 mg/m2 IV weekly for 12 continuous weeks, trastuzumab 6 mg/kg IV (with initial 8-mg/kg IV loading dose) Q3W for 4 cycles & pertuzumab 420 mg IV (with initial 840-mg IV loading dose) Q3W for 4 cycles. During adjuvant phase, participants will continue to receive following study treatments Q3W to complete up to 1 year HER2-target therapy inclusive of therapy given both in neoadjuvant & adjuvant setting: placebo 1200 mg IV Q3W, trastuzumab 6 mg/kg IV (with initial 8-mg/kg IV loading dose) Q3W, & pertuzumab 420 mg IV (with initial 840-mg IV loading dose) Q3W. Participants who do not achieve pCR have option of receiving blinded atezolizumab + trastuzumab emtansine post surgery for 14 cycles. In response to USM DIL, dated 3 Feb 2021 treatment with placebo must be discontinued.
  Interventions: Drug: Placebo; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel; Drug: Trastuzumab; Drug: Pertuzumab; Drug: Trastuzumab Emtansine

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered as per the schedule specified in the respective arm.
  Other Names: Tecentriq
  Arms: Atezolizumab +ddAC-PacHP
Drug: Placebo — Placebo matched to atezolizumab will be administered as per the schedule specified in the respective arm.
  Arms: Placebo + ddAC-PacHP
Drug: Doxorubicin — Doxorubicin will be administered as per the schedule specified in the respective arm.
  Other Names: Adriamycin
Drug: Cyclophosphamide — Cyclophosphamide will be administered as per the schedule specified in the respective arm.
  Other Names: Cytoxan; Neosar
Drug: Paclitaxel — Paclitaxel will be administered as per the schedule specified in the respective arm.
  Other Names: Taxol
Drug: Trastuzumab — Trastuzumab will be administered as per the schedule specified in the respective arm.
  Other Names: Herceptin
Drug: Pertuzumab — Pertuzumab will be administered as per the schedule specified in the respective arm.
  Other Names: Perjeta
Drug: Trastuzumab Emtansine — Participants without pCR have the option of receiving adjuvant atezolizumab/placebo combined with Trastuzumab Emtansine 3.6 mg/kg IV Q3W.
  Other Names: Kadcyla

SUMMARY:
This study (also known as IMpassion050) will evaluate the efficacy and safety of atezolizumab compared with placebo when given in combination with neoadjuvant dose-dense anthracycline (doxorubicin) + cyclophosphamide followed by paclitaxel + trastuzumab + pertuzumab (ddAC-PacHP) in patients with early HER2-positive breast cancer (T2-4, N1-3, M0).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of HER2-positive breast cancer, and hormonal and PD-L1 status, as documented through central testing of a representative tumor tissue specimen
* Primary breast tumor size of > 2 cm by any radiographic measurement
* Stage at presentation: T2-T4, N1-N3, M0 as determined by AJCC staging system, 8th edition
* Pathologic confirmation of nodal involvement with malignancy must be determined by fine needle aspiration or core-needle biopsy. Surgical excision of lymph nodes is not permitted.
* Patients with multifocal tumors are eligible provided at least one focus is sampled and centrally confirmed as HER2-positive.
* Patients with multicentric tumors are eligible provided all discrete lesions are sampled and centrally confirmed as HER2-positive.
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Baseline LVEF >= 55% measured by echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scans
* Adequate hematologic and end-organ function obtained within 14 days prior to initiation of study treatment
* For women of childbearing potential: agreement to remain abstinent or use contraceptive methods, and agreement to refrain from donating eggs
* For men: agreement to remain abstinent or use contraceptive measures, and agreement to refrain from donating sperm

Exclusion Criteria:

* Prior history of invasive breast cancer
* Stage IV (metastatic) breast cancer
* Patients with synchronous bilateral invasive breast cancer
* Prior systemic therapy for treatment of breast cancer
* Previous therapy with anthracyclines or taxanes for any malignancy
* Ulcerating or inflammatory breast cancer
* Undergone incisional and/or excisional biopsy of primary tumor and/or axillary lymph nodes
* Sentinel lymph node procedure or axillary lymph node dissection prior to initiation of neoadjuvant therapy
* History of other malignancy within 5 years prior to screening, with the exception of those patients who have a negligible risk of metastasis or death
* Cardiopulmonary dysfunction
* Dyspnea at rest
* Active or history of autoimmune disease or immune deficiency
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the final dose of atezolizumab/placebo, 6 months after the final dose of doxorubicin, 12 months after the final dose of cyclophosphamide, 6 months after the final dose of paclitaxel, or 7 months after the final dose of trastuzumab, pertuzumab, or trastuzumab emtansine whichever occurs last

Exclusion Criteria Related to Trastuzumab Emtansine in the Adjuvant Setting:

* Patients who achieved pCR
* Evidence of clinically evident gross residual or recurrent disease following neoadjuvant therapy and surgery
* Unable to complete surgery with curative intent after conclusion of neoadjuvant systemic therapy
* Patient discontinued treatment with trastuzumab because of toxicity during the neoadjuvant phase of the study
* Clinically significant history of liver disease, including cirrhosis, current alcohol abuse, autoimmune hepatic disorders, or sclerosis cholangitis
* Patients with Grade >=2 peripheral neuropathy
* Prior treatment with trastuzumab emtansine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2023-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (76):
- United States (3):
  - HCA Midwest Division, Kansas City, Missouri
  - New York University Medical Center PRIME; NYU Langone Medical Center, New York, New York
  - Tennessee Oncology - Nashville, Nashville, Tennessee
- Brazil (5):
  - Hospital Sao Rafael - HSR, Salvador, Estado de Bahia
  - Hospital Araujo Jorge; Departamento de Ginecologia E Mama, Goiânia, Goiás
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital Perola Byington, São Paulo, São Paulo
- Canada (4):
  - Tom Baker Cancer Centre-Calgary, Calgary, Alberta
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Jewish General Hospital, Montreal, Quebec
  - Hopital du Saint Sacrement, Québec, Quebec
- Czechia (2):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Olomouc; Onkologicka klinika, Olomouc
- Germany (8):
  - Klinikum Essen-Mitte Ev. Huyssens-Stiftung / Knappschafts GmbH; Klinik für Senologie / Brustzentrum, Essen
  - Praxis für Interdisziplinäre Onkologie und Hämatologie GbR, Freiburg im Breisgau
  - Kooperatives Mammazentrum Hamburg Krankenhaus Jerusalem, Hamburg
  - Sankt Elisabeth Krankenhaus; Gynaekology, Leipzig
  - Rotkreuzklinikum München; Frauenklinik, München
  - Universitätsklinikum Münster; Klinik für Frauenheilkunde und Geburtshilfe, Münster
  - St. Vincenz-Krankenhaus Paderborn; Haus 3 Frauenklinik, Paderborn
  - Universitätsfrauenklinik Ulm; Abteilung Gynäkologie, Ulm
- Italy (9):
  - Istituto Nazionale Tumori Irccs Fondazione g. PASCALE;U.O.C. Oncologia Medica Senologica, Napoli, Campania
  - Università degli Studi Federico II; Clinica di Oncologia Medica, Napoli, Campania
  - Irccs Centro Di Riferimento Oncologico (CRO); Dipartimento Di Oncologia Medica, Aviano, Friuli Venezia Giulia
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - ASST DEGLI SPEDALI CIVILI DI BRESCIA; Oncologia Medica, Brescia, Lombardy
  - ASST DI MONZA; Oncologia Medica, Monza, Lombardy
  - Istituto Clinico Humanitas;U.O. Oncologia Medica Ed Ematologia, Rozzano, Lombardy
  - Fondazione Del Piemonte Per L'oncologia Ircc Di Candiolo; Dipartimento Oncologico, Candiolo, Piedmont
  - IOV - Istituto Oncologico Veneto - IRCCS; Oncologia Medica II, Padua, Veneto
- Japan (13):
  - National Hospital Organization Shikoku Cancer Center, Ehime
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Hiroshima University Hospital, Hiroshima
  - National Hospital Organization Hokkaido Cancer Center, Hokkaido
  - Hyogo Cancer Center, Hyōgo
  - Kanagawa Cancer Center, Kanagawa
  - Tokai University Hospital, Kanagawa
  - Kumamoto Shinto General Hospital, Kumamoto
  - Fukushima Medical University Hospital, Miyagi
  - Niigata Cancer Center Hospital, Niigata
  - Saitama Medical University International Medical Center, Saitama
  - Toranomon Hospital, Tokyo
  - Showa University Hospital, Tokyo
- Poland (5):
  - Instytut "Centrum Zdrowia Matki Polki"; Klinika Onkologii, ?ód?
  - Narodowy Inst.Onkol.im.Sklodowskiej-Curie Panstw.Inst.Bad Gliwice; Centr.Diagn.i Lecz.Chor.Piersi, Gliwice
  - Regionalny Szpital Specjalistyczny im. W. Bieganskiego; Oddzial Onkologii Klinicznej, Grudzi?dz
  - Szpital Uniwersytecki w Krakowie, Oddzia? Kliniczny Kliniki Onkologii, Krakow
  - Narodowy Inst.Onkologii im.Sklodowskiej-Curie Panstw.Inst.Bad; Klinika Nowtw.Piersi i Chir.Rekonstr, Warsaw
- Russia (6):
  - FSBI National Medical Research Radiological Center; A. TSYB MEDICAL RADIOLOGICAL RESEARCH CENTER, Obninsk, Kaluga Oblast
  - City Clinical Oncology Hospital, Moscow, Moscow Oblast
  - SBIH "Moscow Clinical Scientific and Practical Center named after A.S. Loginov of DHM", Moskva, Moscow Oblast
  - Blokhin Cancer Research Center; Combined Treatment, Moskva, Moscow Oblast
  - Republican Clinical Oncology Dispensary of Ministry of Healthcare of Tatarstan Republic, Kazan', Tatarstan Republic
  - Petrov Research Inst. of Oncology, Saint Petersburg
- South Korea (4):
  - Gachon University Gil Medical Center, Incheon
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Samsung Medical Centre; Oncology, Seoul
- Spain (13):
  - Hospital Universitari Germans Trias i Pujol; Servicio de Oncologia, Badalona, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Sant Andreu de la Barca, Barcelona
  - Hospital Universitario Virgen de La Arrixaca; Servicio De Oncologia, El Palmar, Murcia
  - Clinica Universitaria de Navarra; Servicio de Oncologia, Pamplona, Navarre
  - Hospital Clínic i Provincial; Servicio de Hematología y Oncología, Barcelona
  - Complejo Asistencial Universitario De Burgos; Servicio de Oncologia, Burgos
  - Hospital Clinico de Granada; Servicio de Oncologia, Granada
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico; Servicio de Oncologia, Jaén
  - Hospital Universitari Arnau de Vilanova de Lleida; Servicio de Oncologia, Lleida
  - Clinica Universidad de Navarra Madrid; Servicio de Oncología, Madrid
  - Centro Integral Oncologico Clara Campal; Servicio de Oncología, Madrid
  - Hospital Universitario Virgen Macarena; Servicio de Oncologia, Seville
  - Hospital Universitario Virgen del Rocio; Servicio de Oncologia, Seville
- Taiwan (4):
  - China Medical University Hospital; Surgery, Taichung
  - Mackay Memorial Hospital; Dept of Surgery, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center; Hemato-Oncology, Taipei
  - Chang Gung Medical Foundation - Linkou; Dept of Surgery, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Huober J, Barrios CH, Niikura N, Jarzab M, Chang YC, Huggins-Puhalla SL, Pedrini J, Zhukova L, Graupner V, Eiger D, Henschel V, Gochitashvili N, Lambertini C, Restuccia E, Zhang H; IMpassion050 Trial Investigators. Atezolizumab With Neoadjuvant Anti-Human Epidermal Growth Factor Receptor 2 Therapy and Chemotherapy in Human Epidermal Growth Factor Receptor 2-Positive Early Breast Cancer: Primary Results of the Randomized Phase III IMpassion050 Trial. J Clin Oncol. 2022 Sep 1;40(25):2946-2956. doi: 10.1200/JCO.21.02772. Epub 2022 Jun 28. PMID 35763704

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 74 centers in 12 countries.
Pre-assignment Details: A total of 669 participants were screened, of which a total of 454 participants were enrolled.
Groups:
- Atezolizumab +ddAC-PacHP: Participants received atezolizumab (atezo) 840 mg IV Q2W for 4 cycles during neoadjuvant phase with ddAC (doxorubicin 60 mg/m2 & cyclophosphamide 600 mg/m2 IV), followed by atezo 1200 mg IV Q3W for 4 cycles with paclitaxel 80 mg/m2 IV weekly for 12 continuous weeks, trastuzumab 6 mg/kg IV (with initial 8mg/kg IV loading dose) Q3W for 4 cycles, & pertuzumab 420 mg IV (with initial 840-mg IV loading dose) Q3W for 4 cycles. During adjuvant phase, participants continued to receive following study treatments Q3W to complete up to 1 year HER2-target therapy inclusive of therapy given both in neoadjuvant and adjuvant setting: atezo 1200 mg IV Q3W, trastuzumab 6 mg/kg IV (with initial 8-mg/kg IV loading dose) Q3W, & pertuzumab 420 mg IV (with initial 840-mg IV loading dose) Q3W. Participants who did not achieve pCR had option of receiving blinded atezo+trastuzumab emtansine post surgery for 14 cycles. In response to USM DIL dated 3 Feb 2021 treatment with atezo was discontinued.
- Placebo + ddAC-PacHP: Participants received placebo 840 mg IV Q2W for 4 cycles during neoadjuvant phase with ddAC (doxorubicin 60 mg/m2 & cyclophosphamide 600 mg/m2 IV), followed by placebo 1200 mg IV Q3W for 4 cycles with paclitaxel 80 mg/m2 IV weekly for 12 continuous weeks, trastuzumab 6 mg/kg IV (with initial 8-mg/kg IV loading dose) Q3W for 4 cycles & pertuzumab 420 mg IV (with initial 840-mg IV loading dose) Q3W for 4 cycles. During adjuvant phase, participants continued to receive following study treatments Q3W to complete up to 1 year HER2-target therapy inclusive of therapy given both in neoadjuvant & adjuvant setting: placebo 1200 mg IV Q3W, trastuzumab 6 mg/kg IV (with initial 8-mg/kg IV loading dose) Q3W, & pertuzumab 420 mg IV (with initial 840-mg IV loading dose) Q3W. Participants who did not achieve pCR had option of receiving blinded atezolizumab + trastuzumab emtansine post surgery for 14 cycles. In response to USM DIL, dated 3 Feb 2021 treatment with placebo was discontinued.
Period: Overall Study
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Started | 226 | 228
Completed | 206 | 205
Not Completed | 20 | 23
Not completed — Death | 11 | 13
Not completed — Physician Decision | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 5 | 6
Not completed — TSH result is unstable | 0 | 1
Not completed — Disease relapse | 1 | 0
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP | Total
Number analyzed (Participants) | 226 | 228 | 454
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.3 (10.7) | 50.8 (10.4) | 50.6 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 225 | 227 | 452
  Male | 1 | 1 | 2
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 26 | 33 | 59
  Not Hispanic or Latino | 195 | 191 | 386
  Not Reported | 5 | 4 | 9
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 62 | 66 | 128
  Black or African American | 8 | 13 | 21
  White | 149 | 142 | 291
  Multiple | 2 | 3 | 5
  Unknown | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pathological Complete Response (pCR) in the PD-L1-Positive Population (IC 1/2/3)
Description: pCR is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (NAST) (i.e., ypT0/is ypN0 in the current American Joint Committee on Cancer [AJCC] staging system, 8th edition). Treatment comparison was made using Cochran-Mantel-Haenszel test stratified by disease stage (T2 vs. T3-4) and hormone receptor status (estrogen receptor (ER) positive and/or progesterone receptor (PgR) positive vs. ER negative and PgR negative).
Time Frame: From randomization to approximately 6 months
Population: The PD-L1-positive population is defined as participants in the Intent-to-Treat (ITT) population whose PD-L1 status is IC1/2/3 at the time of randomization.
Measure: Number; unit: Percentage of Participants
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Number analyzed (Participants) | 109 | 109
Percentage of Participants | 64.2 [54.47 to 73.17] | 72.5 [63.10 to 80.60]
Statistical Analysis 1: Comparison: Atezolizumab +ddAC-PacHP vs Placebo + ddAC-PacHP; Test type: Superiority; p = 0.1846, Cochran-Mantel-Haenszel — The threshold for statistical significance was a p-value =0.048; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.37 to 1.21]

2. Primary Outcome: pCR in the ITT Population
Description: pCR is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (NAST) (i.e., ypT0/is ypN0 in the current American Joint Committee on Cancer [AJCC] staging system, 8th edition). Treatment comparison was made using Cochran-Mantel-Haenszel test stratified by disease stage (T2 vs. T3-4) and hormone receptor status (ER positive and/or PgR positive vs. ER negative and PgR negative).
Time Frame: From randomization to approximately 6 months
Population: The ITT population is defined as all randomized participants, regardless of whether the assigned study treatment was received.
Measure: Number; unit: Percentage of Participants
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Number analyzed (Participants) | 226 | 228
Percentage of Participants | 62.4 [55.72 to 68.73] | 62.7 [56.09 to 69.01]
Statistical Analysis 1: Comparison: Atezolizumab +ddAC-PacHP vs Placebo + ddAC-PacHP; Test type: Superiority; p = 0.9551, Cochran-Mantel-Haenszel — The threshold for statistical significance was a p-value =0.002; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.67 to 1.46]

3. Secondary Outcome: Percentage of Participants With pCR Based on Hormone Receptor Status
Description: pCR (ypT0/is ypN0) based upon hormone receptor status (estrogen receptor [ER]/progesterone receptor [PgR] positive or ER/PgR negative).
Time Frame: From randomization to approximately 24 months
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Number analyzed (Participants) | 226 | 228
Percentage of Participants
  ER+ and/or PgR+: number analyzed (Participants) | 116 | 117
  ER+ and/or PgR+ | 50.9 | 54.7
  ER- and/or PgR-: number analyzed (Participants) | 110 | 111
  ER- and/or PgR- | 74.5 | 71.2

4. Secondary Outcome: Percentage of Participants With pCR in the PD-L1-Negative Population
Description: pCR (ypT0/is ypN0) in the IC 0 Population
Time Frame: From randomization to approximately 24 months
Population: The PD-L1-negative population is defined as participants in the ITT population whose PD-L1 status is IC 0 at the time of randomization.
Measure: Number; unit: Percentage of Participants
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Number analyzed (Participants) | 117 | 119
Percentage of Participants | 60.7 [51.23 to 69.59] | 53.8 [44.41 to 62.96]

5. Secondary Outcome: Event-Free Survival (EFS)
Description: EFS defined as the time from randomization to the first documented disease recurrence, unequivocal tumor progression determined by the treating investigator, or death from any cause, whichever occurs first, in all patients and based upon hormone receptor status (ER/PgR positive or ER/PgR negative) and PD-L1 status (IC 0; IC 1/2/3).
Time Frame: From randomization to first documented disease recurrence, unequivocal tumor progression determined by the treating investigator, or death from any cause (up to approximately 54 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Number analyzed (Participants) | 226 | 228
Months
  All Participants | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached
  PD-L1 IC1/2/3 Participants: number analyzed (Participants) | 109 | 109
  PD-L1 IC1/2/3 Participants | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached.
  PD-L1 IC0 Participants: number analyzed (Participants) | 117 | 119
  PD-L1 IC0 Participants | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached
  ER/PgR Negative Participants: number analyzed (Participants) | 110 | 111
  ER/PgR Negative Participants | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached
  ER/PgR Positive Participants: number analyzed (Participants) | 116 | 117
  ER/PgR Positive Participants | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached
Statistical Analysis 1: Comparison: Atezolizumab +ddAC-PacHP vs Placebo + ddAC-PacHP; All Participants; Test type: Superiority; Log Rank; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.50 to 1.59]
Statistical Analysis 2: Comparison: Atezolizumab +ddAC-PacHP vs Placebo + ddAC-PacHP; PD-L1 IC1/2/3; Test type: Superiority; Log Rank; Hazard Ratio (HR) = 1.67, 95% CI 2-sided [0.65 to 4.32]
Statistical Analysis 3: Comparison: Atezolizumab +ddAC-PacHP vs Placebo + ddAC-PacHP; PD-L1 IC0 Participants; Test type: Superiority; Log Rank; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.27 to 1.22]
Statistical Analysis 4: Comparison: Atezolizumab +ddAC-PacHP vs Placebo + ddAC-PacHP; ER/PgR Negative Participants; Test type: Superiority; Log Rank; Hazard Ratio (HR) = 1.28, 95% CI 2-sided [0.58 to 2.82]
Statistical Analysis 5: Comparison: Atezolizumab +ddAC-PacHP vs Placebo + ddAC-PacHP; ER/PgR Positive Participants; Test type: Superiority; Log Rank; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.24 to 1.36]

6. Secondary Outcome: Disease-Free Survival (DFS)
Description: DFS defined as the time from surgery to the first documented disease recurrence or death from any cause, whichever occurs first, in all patients who undergo surgery and based upon PD-L1 status (IC 0; IC 1/2/3).
Time Frame: Time from surgery to first documented disease recurrence or death from any cause (up to approximately 54 months)
Population: The DFS-evaluable population is defined as participants in the ITT population who undergo surgery.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Number analyzed (Participants) | 217 | 217
Months
  All Participants | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached
  PD-L1 IC1/2/3: number analyzed (Participants) | 104 | 106
  PD-L1 IC1/2/3 | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached
  PD-L1 IC0: number analyzed (Participants) | 113 | 111
  PD-L1 IC0 | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached
Statistical Analysis 1: Comparison: Atezolizumab +ddAC-PacHP vs Placebo + ddAC-PacHP; All Participants; Test type: Superiority; Log Rank; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.38 to 1.32]
Statistical Analysis 2: Comparison: Atezolizumab +ddAC-PacHP vs Placebo + ddAC-PacHP; PD-L1 IC1/2/3; Test type: Superiority; Log Rank; Hazard Ratio (HR) = 1.38, 95% CI 2-sided [0.51 to 3.69]
Statistical Analysis 3: Comparison: Atezolizumab +ddAC-PacHP vs Placebo + ddAC-PacHP; PD-L1 IC0; Test type: Superiority; Log Rank; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.19 to 1.02]

7. Secondary Outcome: Overall Survival (OS)
Description: OS defined as the time from randomization to death from any cause in all participants and based upon PD-L1 status (IC 0; IC 1/2/3).
Time Frame: From randomization to date of death from any cause (up to approximately 54 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Number analyzed (Participants) | 226 | 228
Months
  All Participants | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached
  PD-L1 IC1/2/3: number analyzed (Participants) | 109 | 109
  PD-L1 IC1/2/3 | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached
  PD-L1 IC0: number analyzed (Participants) | 117 | 119
  PD-L1 IC0 | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached | NA [NA to NA] — The median time to event based on Kaplan-Meier estimates was not reached
Statistical Analysis 1: Comparison: Atezolizumab +ddAC-PacHP vs Placebo + ddAC-PacHP; All Participants; Test type: Superiority; Log Rank; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.40 to 2.00]
Statistical Analysis 2: Comparison: Atezolizumab +ddAC-PacHP vs Placebo + ddAC-PacHP; PD-L1 IC1/2/3; Test type: Superiority; Log Rank; Hazard Ratio (HR) = 1.75, 95% CI 2-sided [0.42 to 7.33]
Statistical Analysis 3: Comparison: Atezolizumab +ddAC-PacHP vs Placebo + ddAC-PacHP; PD-L1 IC0; Test type: Superiority; Log Rank; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.21 to 1.59]

8. Secondary Outcome: Mean Changes From Baseline in Function (Role, Physical)
Description: EORTC QLQ-C30 is a self-reported questionnaire that included functional scales (physical, role, cognitive, emotional, social), symptom scales (fatigue, pain, nausea/vomiting), global health scale/quality of life (GHS/QOL) and single items (dyspnea, appetite loss, insomnia, constipation, diarrhea, financial difficulties). Questions 1-28 on the QLQ-C30 were on a 4-point scale (1=Not at All to 4=Very Much). Questions 29-30 (GHS scale) were on a 7-point scale (1=Very Poor to 7=Excellent). For this instrument, GHS/QOL and functional scales were linearly transformed so each score ranged 0-100, where lower scores indicate poorer functioning (e.g., worsening) and higher scores indicate better functioning (e.g., improvement).
Time Frame: Baseline; Day 1 of Cycle 1-9, on Day 1 of every other cycle thereafter until Cycle 22; at the treatment discontinuation or early termination visit and follow up visit. Cycle 1-4, each cycle is 14 days. Cycle 5-22, each cycle is 21 days.
Population: The patient-reported outcomes (PRO)-evaluable population is defined as participants in the ITT population with a baseline and at least 1 post-baseline PRO assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Number analyzed (Participants) | 223 | 224
Units on a scale
  Role: Baseline | 91.70 (16.28) | 90.85 (20.26)
  Role: Cycle (C) 2 Day (D) 1: number analyzed (Participants) | 222 | 222
  Role: Cycle (C) 2 Day (D) 1 | -13.06 (23.02) | -9.83 (23.08)
  Role: C3D1: number analyzed (Participants) | 219 | 220
  Role: C3D1 | -17.88 (26.20) | -15.15 (22.64)
  Role: C4D1: number analyzed (Participants) | 217 | 216
  Role: C4D1 | -22.27 (27.04) | -17.98 (25.10)
  Role: C5D1: number analyzed (Participants) | 218 | 219
  Role: C5D1 | -24.08 (28.21) | -19.79 (26.36)
  Role: C6D1: number analyzed (Participants) | 215 | 216
  Role: C6D1 | -20.70 (25.46) | -18.60 (25.01)
  Role: C7D1: number analyzed (Participants) | 210 | 210
  Role: C7D1 | -19.21 (25.50) | -16.67 (26.34)
  Role: C8D1: number analyzed (Participants) | 211 | 208
  Role: C8D1 | -21.25 (26.48) | -17.79 (26.39)
  Role: Adjuvant Week 1 D1: number analyzed (Participants) | 206 | 202
  Role: Adjuvant Week 1 D1 | -22.82 (26.70) | -26.24 (31.27)
  Role: Adjuvant Week 7 D43: number analyzed (Participants) | 183 | 176
  Role: Adjuvant Week 7 D43 | -15.48 (22.31) | -15.15 (26.50)
  Role: Adjuvant Week 13 D85: number analyzed (Participants) | 171 | 163
  Role: Adjuvant Week 13 D85 | -14.42 (23.77) | -15.24 (26.99)
  Role: Adjuvant Week 19 D127: number analyzed (Participants) | 155 | 147
  Role: Adjuvant Week 19 D127 | -14.30 (24.26) | -15.42 (25.74)
  Role: Adjuvant Week 25 D169: number analyzed (Participants) | 134 | 127
  Role: Adjuvant Week 25 D169 | -13.68 (24.00) | -15.88 (22.99)
  Role: Adjuvant Week 31 D211: number analyzed (Participants) | 112 | 110
  Role: Adjuvant Week 31 D211 | -13.24 (23.69) | -14.55 (24.43)
  Role: Adjuvant Week 37 D253: number analyzed (Participants) | 91 | 94
  Role: Adjuvant Week 37 D253 | -9.34 (21.11) | -15.43 (27.35)
  Role: End of Treatment (EOT): number analyzed (Participants) | 108 | 116
  Role: End of Treatment (EOT) | -14.04 (25.18) | -18.10 (29.04)
  Role: Follow-Up (FU) 1 D1: number analyzed (Participants) | 62 | 68
  Role: Follow-Up (FU) 1 D1 | -11.02 (25.06) | -17.16 (23.21)
  Role: FU2D92: number analyzed (Participants) | 20 | 33
  Role: FU2D92 | -9.17 (23.24) | -14.65 (25.94)
  Role: FU3D183: number analyzed (Participants) | 3 | 8
  Role: FU3D183 | -16.67 (16.67) | -10.42 (21.71)
  Role: FU4D274: number analyzed (Participants) | 3 | 6
  Role: FU4D274 | -27.78 (25.46) | -25.00 (9.13)
  Role: FU5D457: number analyzed (Participants) | 0 | 1
  Role: FU5D457 |  | -33.33 (NA) — Standard deviation (SD) was non-estimable as only 1 participant was evaluated for this category.
  Physical: Baseline | 92.74 (11.60) | 92.20 (12.92)
  Physical: C2D1: number analyzed (Participants) | 222 | 221
  Physical: C2D1 | -4.32 (9.75) | -3.88 (13.44)
  Physical: C3D1: number analyzed (Participants) | 219 | 220
  Physical: C3D1 | -6.82 (13.39) | -7.18 (12.91)
  Physical: C4D1: number analyzed (Participants) | 217 | 216
  Physical: C4D1 | -11.98 (17.67) | -9.48 (14.65)
  Physical: C5D1: number analyzed (Participants) | 218 | 219
  Physical: C5D1 | -12.84 (16.76) | -10.67 (15.91)
  Physical: C6D1: number analyzed (Participants) | 215 | 216
  Physical: C6D1 | -12.25 (15.97) | -11.40 (17.05)
  Physical: C7D1: number analyzed (Participants) | 210 | 210
  Physical: C7D1 | -11.33 (14.86) | -11.45 (17.43)
  Physical: C8D1: number analyzed (Participants) | 211 | 208
  Physical: C8D1 | -13.30 (17.11) | -11.56 (17.54)
  Physical: Adjuvant Week 1 D1: number analyzed (Participants) | 206 | 202
  Physical: Adjuvant Week 1 D1 | -12.27 (18.26) | -12.19 (19.27)
  Physical: Adjuvant Week 7 D43: number analyzed (Participants) | 183 | 176
  Physical: Adjuvant Week 7 D43 | -8.96 (14.74) | -8.60 (16.33)
  Physical: Adjuvant Week 13 D85: number analyzed (Participants) | 171 | 163
  Physical: Adjuvant Week 13 D85 | -8.38 (14.97) | -8.88 (15.04)
  Physical: Adjuvant Week 19 D127: number analyzed (Participants) | 154 | 147
  Physical: Adjuvant Week 19 D127 | -9.22 (15.17) | -10.03 (15.52)
  Physical: Adjuvant Week 25 D169: number analyzed (Participants) | 134 | 127
  Physical: Adjuvant Week 25 D169 | -9.35 (16.19) | -8.45 (14.34)
  Physical: Adjuvant Week 31 D211: number analyzed (Participants) | 112 | 110
  Physical: Adjuvant Week 31 D211 | -7.80 (13.69) | -9.88 (15.84)
  Physical: Adjuvant Week 37 D253: number analyzed (Participants) | 91 | 94
  Physical: Adjuvant Week 37 D253 | -7.77 (13.67) | -10.78 (16.82)
  Physical: EOT: number analyzed (Participants) | 109 | 116
  Physical: EOT | -8.20 (15.78) | -13.05 (19.17)
  Physical: FU1D1: number analyzed (Participants) | 62 | 68
  Physical: FU1D1 | -8.06 (18.11) | -11.57 (19.29)
  Physical: FU2D92: number analyzed (Participants) | 20 | 33
  Physical: FU2D92 | -3.33 (12.52) | -9.90 (15.73)
  Physical: FU3D183: number analyzed (Participants) | 3 | 8
  Physical: FU3D183 | 2.22 (16.78) | -14.17 (7.51)
  Physical: FU4D274: number analyzed (Participants) | 3 | 6
  Physical: FU4D274 | 0.00 (20.00) | -6.67 (11.93)
  Physical: FU5D457: number analyzed (Participants) | 0 | 1
  Physical: FU5D457 |  | 60.00 (NA) — SD was non-estimable as only 1 participant was evaluated for this category.

9. Secondary Outcome: Mean Changes From Baseline in Global Health Status
Description: EORTC QLQ-C30 is a self-reported questionnaire that included functional scales (physical, role, cognitive, emotional, social), symptom scales (fatigue, pain, nausea/vomiting), GHS/QOL and single items (dyspnea, appetite loss, insomnia, constipation, diarrhea, financial difficulties). Questions 1-28 on the QLQ-C30 were on a 4-point scale (1=Not at All to 4=Very Much). Questions 29-30 (GHS scale) were on a 7-point scale (1=Very Poor to 7=Excellent). For this instrument, GHS/QOL and functional scales were linearly transformed so each score ranged 0-100, where lower scores indicate poorer functioning (e.g., worsening) and higher scores indicate better functioning (e.g., improvement).
Time Frame: as for outcome 8
Population: The PRO-evaluable population is defined as participants in the ITT population with a baseline and at least 1 post-baseline PRO assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Number analyzed (Participants) | 223 | 224
Units on a scale
  Baseline | 76.49 (19.33) | 76.79 (19.05)
  C2D1: number analyzed (Participants) | 222 | 222
  C2D1 | -7.28 (19.70) | -6.31 (19.54)
  C3D1: number analyzed (Participants) | 219 | 220
  C3D1 | -10.96 (22.16) | -8.33 (20.93)
  C4D1: number analyzed (Participants) | 217 | 216
  C4D1 | -13.67 (22.47) | -10.88 (21.51)
  C5D1: number analyzed (Participants) | 218 | 219
  C5D1 | -14.14 (23.76) | -12.63 (23.66)
  C6D1: number analyzed (Participants) | 215 | 216
  C6D1 | -12.33 (22.10) | -9.99 (20.96)
  C7D1: number analyzed (Participants) | 210 | 210
  C7D1 | -11.47 (19.81) | -10.52 (21.59)
  C8D1: number analyzed (Participants) | 211 | 208
  C8D1 | -12.72 (22.45) | -10.86 (22.66)
  Adjuvant Week 1 D1: number analyzed (Participants) | 206 | 202
  Adjuvant Week 1 D1 | -7.89 (21.89) | -7.14 (23.68)
  Adjuvant Week 7 D43: number analyzed (Participants) | 183 | 176
  Adjuvant Week 7 D43 | -7.51 (22.97) | -5.21 (21.96)
  Adjuvant Week 13 D85: number analyzed (Participants) | 171 | 163
  Adjuvant Week 13 D85 | -7.07 (22.31) | -6.75 (21.13)
  Adjuvant Week 19 D127: number analyzed (Participants) | 155 | 147
  Adjuvant Week 19 D127 | -7.20 (21.47) | -6.01 (20.52)
  Adjuvant Week 25 D169: number analyzed (Participants) | 134 | 127
  Adjuvant Week 25 D169 | -8.02 (21.10) | -5.05 (20.39)
  Adjuvant Week 31 D211: number analyzed (Participants) | 112 | 110
  Adjuvant Week 31 D211 | -7.29 (21.75) | -7.80 (22.56)
  Adjuvant Week 37 D253: number analyzed (Participants) | 91 | 94
  Adjuvant Week 37 D253 | -5.95 (21.71) | -6.03 (20.72)
  EOT: number analyzed (Participants) | 109 | 116
  EOT | -5.96 (22.08) | -9.41 (24.29)
  FU1D1: number analyzed (Participants) | 62 | 68
  FU1D1 | -3.90 (21.64) | -5.15 (21.01)
  FU2D92: number analyzed (Participants) | 20 | 33
  FU2D92 | -1.25 (19.55) | -3.03 (16.11)
  FU3D183: number analyzed (Participants) | 3 | 8
  FU3D183 | -8.33 (8.33) | -7.29 (15.06)
  FU4D274: number analyzed (Participants) | 3 | 6
  FU4D274 | -13.89 (12.73) | -31.94 (37.42)
  FU5D457: number analyzed (Participants) | 0 | 1
  FU5D457 |  | -16.67 (NA) — SD was non-estimable as only 1 participant was evaluated for this category.

10. Secondary Outcome: Percentage of Participants With Adverse Events
Time Frame: From randomization up end of study (approximately 4 years and 7 months)
Population: The safety-evaluable population is defined as participants who received at least one dose of any study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Number analyzed (Participants) | 226 | 225
Percentage of Participants | 100 | 100

11. Secondary Outcome: Maximum Serum Concentration (Cmax) of Atezolizumab
Description: Cmax is the maximum (or peak) concentration that a study drug achieves in the body.
Time Frame: 30 minutes post infusion on Day 1 Cycle (C) 1.
Population: The pharmacokinetic (PK)-evaluable population is defined as all participants who received any dose of study medication and who have at least one post-baseline PK sample available.
Measure: Mean (Standard Deviation); unit: micrograms/milliliters (ug/mL)
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Number analyzed (Participants) | 219 | 0
micrograms/milliliters (ug/mL) | 348 (122) |

12. Secondary Outcome: Minimum Serum Concentration (Cmin) of Atezolizumab
Description: Cmin is the minimum (or trough) concentration that a study drug achieves in the body.
Time Frame: Pre-dose on Day 1 Cycle (C) 2, 3, 4, 8, 12, 16, ATDV (an average of 1 year). C 2-4, each C is 14 days. C 8-16, each C is 21 days. With protocol version 5, collection is only required ATDV/completion (an average of 1 year).
Population: The PK-evaluable population is defined as all participants who received any dose of study medication and who have at least one post-baseline PK sample available.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Number analyzed (Participants) | 226 | 0
ug/mL
  C2D1/predose: number analyzed (Participants) | 222 | 0
  C2D1/predose | 103 (40.3) |
  C3D1/predose: number analyzed (Participants) | 214 | 0
  C3D1/predose | 163 (44.4) |
  C4D1/predose: number analyzed (Participants) | 212 | 0
  C4D1/predose | 204 (51.9) |
  C8D1/predose: number analyzed (Participants) | 203 | 0
  C8D1/predose | 225 (97.1) |
  C12D1/predose: number analyzed (Participants) | 166 | 0
  C12D1/predose | 217 (101) |
  C16D1/predose: number analyzed (Participants) | 133 | 0
  C16D1/predose | 226 (114) |

13. Secondary Outcome: Trough Concentration (Ctrough) for Pertuzumab and Trastuzumab in Serum
Time Frame: Pre-dose on Day 1 Cycle (C) 8, 12, and at treatment discontinuation visit (ATDV) (an average of 1 year). C 1-4, each C is 14 days. C 8-12, each C is 21 days. With protocol version 5, collection is only required ATDV/completion (an average of 1 year).
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Number analyzed (Participants) | 226 | 225
ug/mL
  Pertuzumab: C8D1/predose: number analyzed (Participants) | 205 | 201
  Pertuzumab: C8D1/predose | 93.2 (40.7) | 94.8 (39.8)
  Pertuzumab: C12D1/predose: number analyzed (Participants) | 150 | 147
  Pertuzumab: C12D1/predose | 87.7 (58.4) | 91.6 (59.7)
  Trastuzumab: C8D1/predose: number analyzed (Participants) | 205 | 201
  Trastuzumab: C8D1/predose | 58.5 (29.1) | 56.5 (23.9)
  Trastuzumab: C12D1/predose: number analyzed (Participants) | 150 | 147
  Trastuzumab: C12D1/predose | 62.4 (32.7) | 60.4 (30.9)

14. Secondary Outcome: Cmax of Trastuzumab Emtansine in Serum
Description: Cmax is the maximum (or peak) concentration that a study drug achieves in the body.
Time Frame: Day 1 of Cycle 9 and Cycle 12, at treatment disontinuation visit (an average of 1 year). Cycle 9 and 12 are each 21 days. With protocol version 5, collection is only required at the time of treatment discontinuation/completion (an average of 1 year).
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Number analyzed (Participants) | 53 | 49
ug/mL
  C9D1: number analyzed (Participants) | 52 | 46
  C9D1 | 84.3 (29.0) | 80.5 (26.8)
  C12D1: number analyzed (Participants) | 49 | 46
  C12D1 | 82.0 (32.2) | 82.0 (37.2)

15. Secondary Outcome: Cmin of Trastuzumab Emtansine in Serum
Description: Cmin is the minimum (or trough) concentration that a study drug achieves in the body.
Time Frame: as for outcome 14
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Number analyzed (Participants) | 53 | 49
ug/mL | 2.18 (5.09) | 1.22 (1.49)

16. Secondary Outcome: Number of Participants With Treatment-Emergent Anti-Drug Antibodies (ADAs) to Atezolizumab
Description: Participants were considered to be treatment-emergent ADA-positive if they were ADA-negative or had missing data at baseline but developed an ADA response following study drug exposure (treatment-induced ADA response), or if they were ADA-positive at baseline and the titer of one or more post-baseline samples was at least 0.60 titer units greater than the titer of the baseline sample (treatment-enhanced ADA response). Participants were considered to be treatment-emergent ADA-negative if they were ADA-negative or were missing data at baseline and all post-baseline samples were negative, or if they were ADA-positive at baseline but did not have any post-baseline samples with a titer that was at least 0.60 titer units greater than the titer of the baseline sample (treatment unaffected).
Time Frame: Day 1 Cycle (C) 1, 2, 3, 4, 8, 12, 16, at treatment discontinuation visit (ATDV) (an average of 1 year). C 1-4, each C is 14 days. C 8-16, each C is 21 days. With protocol version 5, collection is only required ATDV/completion (an average of 1 year).
Population: The immunogenicity analysis included all safety evealuable participants who had at least one baseline or post-baseline ADA result from at least one sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Number analyzed (Participants) | 225 | 0
Participants
  Baseline (BL): ADA Positive | 1 |
  BL: ADA Negative | 224 |
  Post-BL: Treatment-Emergent ADA Positive | 7 |
  Post-BL: Treatment-Emergent ADA Negative | 218 |

17. Secondary Outcome: Number of Participants With Treatment-Emergent ADAs to Trastuzumab
Description: as for outcome 16
Time Frame: Day 1 Cycle (C) 1, 8, 12 and at treatment discontinuation visit (ATDV) (an average of 1 year). C 1-4, each C is 14 days. C 8-12, each C is 21 days. With protocol version 5, collection is only required ATDV/completion (an average of 1 year).
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Number analyzed (Participants) | 226 | 225
Participants
  BL: ADA Positive: number analyzed (Participants) | 216 | 207
  BL: ADA Positive | 2 | 1
  BL: ADA Negative: number analyzed (Participants) | 216 | 207
  BL: ADA Negative | 214 | 206
  Post-BL: Treatment-Emergent ADA Positive: number analyzed (Participants) | 213 | 216
  Post-BL: Treatment-Emergent ADA Positive | 1 | 0
  Post-BL: Treatment-Emergent ADA Negative: number analyzed (Participants) | 213 | 216
  Post-BL: Treatment-Emergent ADA Negative | 212 | 216

18. Secondary Outcome: Number of Participants With Treatment-Emergent ADAs to Pertuzumab
Description: as for outcome 16
Time Frame: Day 1 of Cycle (C) 1, 8, 12, and at treatment discontinuation visit (ATDV) (an average of 1 year). C 1-4, each C is 14 days. C 8-12, each C is 21 days. With protocol version 5, collection is only required ATDV/completion (an average of 1 year).
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Number analyzed (Participants) | 226 | 225
Participants
  BL: ADA Positive: number analyzed (Participants) | 216 | 209
  BL: ADA Positive | 6 | 3
  BL: ADA Negative: number analyzed (Participants) | 216 | 209
  BL: ADA Negative | 210 | 206
  Post-BL: Treatment-Emergent ADA Positive: number analyzed (Participants) | 213 | 217
  Post-BL: Treatment-Emergent ADA Positive | 4 | 3
  Post-BL: Treatment-Emergent ADA Negative: number analyzed (Participants) | 213 | 217
  Post-BL: Treatment-Emergent ADA Negative | 209 | 214

19. Secondary Outcome: Number of Participants With Treatment-Emergent ADAs to Trastuzumab Emtansine
Description: as for outcome 16
Time Frame: as for outcome 14
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Number analyzed (Participants) | 57 | 55
Participants
  BL: ADA Positive: number analyzed (Participants) | 52 | 50
  BL: ADA Positive | 3 | 2
  BL: ADA Negative: number analyzed (Participants) | 52 | 50
  BL: ADA Negative | 49 | 48
  Post-BL: Treatment-Emergent ADA Positive | 1 | 1
  Post-BL: Treatment-Emergent ADA Negative | 56 | 54

20. Secondary Outcome: Percentage of Participants With pCR Based on PIK3CA Mutation Status
Description: pCR is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (NAST) (i.e., ypT0/is ypN0 in the current American Joint Committee on Cancer [AJCC] staging system, 8th edition).
Time Frame: From randomization to approximately 24 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Number analyzed (Participants) | 226 | 228
Participants
  Mutated: number analyzed (Participants) | 67 | 61
  Mutated | 40 | 34
  Wildtype: number analyzed (Participants) | 150 | 155
  Wildtype | 98 | 101
  Missing: number analyzed (Participants) | 9 | 12
  Missing | 3 | 8

21. Secondary Outcome: EFS Based on PIK3CA Mutation Status
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Number analyzed (Participants) | 226 | 228
Months
  Missing: number analyzed (Participants) | 9 | 12
  Missing | NA [NA to NA] — Too few events to calculate the median and 95% confidence intervals. | NA [NA to NA] — Too few events to calculate the median and 95% confidence intervals.
  Mutated: number analyzed (Participants) | 67 | 61
  Mutated | NA [NA to NA] — Too few events to calculate the median and 95% confidence intervals. | NA [NA to NA] — Too few events to calculate the median and 95% confidence intervals.
  Wildtype: number analyzed (Participants) | 150 | 155
  Wildtype | NA [NA to NA] — Too few events to calculate the median and 95% confidence intervals. | NA [NA to NA] — Too few events to calculate the median and 95% confidence intervals.
Statistical Analysis 1: Comparison: Atezolizumab +ddAC-PacHP vs Placebo + ddAC-PacHP; PIK3CA-Missing; Test type: Superiority; Regression, Cox; Hazard Ratio (HR) = 2.38, 95% CI 2-sided [0.22 to 26.42]
Statistical Analysis 2: Comparison: Atezolizumab +ddAC-PacHP vs Placebo + ddAC-PacHP; PIK3CA-Mutated; Test type: Superiority; Regression, Cox; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.23 to 1.90]
Statistical Analysis 3: Comparison: Atezolizumab +ddAC-PacHP vs Placebo + ddAC-PacHP; PIK3CA-Wildtype; Test type: Superiority; Regression, Cox; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.45 to 1.87]

22. Secondary Outcome: DFS Based on PIK3CA Mutation Status
Time Frame: Time from surgery to first documented disease recurrence or death from any cause (up to approximately 54 months)
Population: The DFS-evaluable population is defined as participants in the ITT population who undergo surgery.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Number analyzed (Participants) | 217 | 217
Months
  Missing: number analyzed (Participants) | 8 | 11
  Missing | NA [NA to NA] — Too few events to calculate the median and 95% confidence intervals. | NA [NA to NA] — Too few events to calculate the median and 95% confidence intervals.
  Mutated: number analyzed (Participants) | 66 | 57
  Mutated | NA [NA to NA] — Too few events to calculate the median and 95% confidence intervals. | NA [NA to NA] — Too few events to calculate the median and 95% confidence intervals.
  Wildtype: number analyzed (Participants) | 143 | 149
  Wildtype | NA [NA to NA] — Too few events to calculate the median and 95% confidence intervals. | NA [NA to NA] — Too few events to calculate the median and 95% confidence intervals.
Statistical Analysis 1: Comparison: Atezolizumab +ddAC-PacHP vs Placebo + ddAC-PacHP; PIK3CA-Missing; Test type: Superiority; Regression, Cox; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.07 to 18.91]
Statistical Analysis 2: Comparison: Atezolizumab +ddAC-PacHP vs Placebo + ddAC-PacHP; PIK3CA-Mutated; Test type: Superiority; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.19 to 1.92]
Statistical Analysis 3: Comparison: Atezolizumab +ddAC-PacHP vs Placebo + ddAC-PacHP; PIK3CA-Wildtype; Test type: Superiority; Regression, Cox; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.33 to 1.55]

23. Secondary Outcome: OS Based on PIK3CA Mutation Status
Time Frame: From randomization to date of death from any cause (up to approximately 54 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
Number analyzed (Participants) | 226 | 228
Months
  Missing: number analyzed (Participants) | 9 | 12
  Missing | NA [NA to NA] — Too few events to calculate the median and 95% confidence intervals. | NA [NA to NA] — Too few events to calculate the median and 95% confidence intervals.
  Mutated: number analyzed (Participants) | 67 | 61
  Mutated | NA [NA to NA] — Too few events to calculate the median and 95% confidence intervals. | NA [NA to NA] — Too few events to calculate the median and 95% confidence intervals.
  Wildtype: number analyzed (Participants) | 150 | 155
  Wildtype | NA [NA to NA] — Too few events to calculate the median and 95% confidence intervals. | NA [NA to NA] — Too few events to calculate the median and 95% confidence intervals.
Statistical Analysis 1: Comparison: Atezolizumab +ddAC-PacHP vs Placebo + ddAC-PacHP; PIK3CA-Missing; Test type: Superiority; Regression, Cox; Hazard Ratio (HR) = 999.99, 95% CI 2-sided [lower limit 0.00] (Upper limit of the CI was not evaluable due to low number of events) — The estimated value is >999.99
Statistical Analysis 2: Comparison: Atezolizumab +ddAC-PacHP vs Placebo + ddAC-PacHP; PIK3CA-Mutated; Test type: Superiority; Regression, Cox; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.10 to 3.53]
Statistical Analysis 3: Comparison: Atezolizumab +ddAC-PacHP vs Placebo + ddAC-PacHP; PIK3CA-Wildtype; Test type: Superiority; Regression, Cox; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.33 to 2.09]

ADVERSE EVENTS:
Time Frame: From randomization up until end of study (approximately 4 years and 7 months)
Description: All-cause mortality was reported based on the Intention-to-Treat (ITT) Population = all randomized participants.
  AEs were recorded for the safety-evaluable population which included all randomized participants who received any dose of study drug.
Arm/Group | Atezolizumab +ddAC-PacHP | Placebo + ddAC-PacHP
All-Cause Mortality (participants affected / at risk) | 11/226 | 13/228
Serious Adverse Events (participants affected / at risk) | 65/226 | 47/225
Other Adverse Events (participants affected / at risk) | 226/226 | 225/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab +ddAC-PacHP (N=226) | Placebo + ddAC-PacHP (N=225)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Aplastic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 10 (12) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (3) | 5 (6)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 4 (4) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 1 (1)
Meibomianitis (Eye disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Immune-mediated pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Capsular contracture associated with breast implant (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 3 (4)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Steatohepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Gastritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Mastitis (Infections and infestations) | 3 (4) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Vascular access site infection (Infections and infestations) | 0 (0) | 2 (2)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0)
Vulval cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Implantation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nervous system neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Meningitis noninfective (Nervous system disorders) | 0 (0) | 1 (1)
Device extrusion (Product Issues) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Adnexal torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Vascular pain (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab +ddAC-PacHP (N=226) | Placebo + ddAC-PacHP (N=225)
Anaemia (Blood and lymphatic system disorders) | 116 (179) | 118 (235)
Leukopenia (Blood and lymphatic system disorders) | 37 (104) | 50 (130)
Lymphopenia (Blood and lymphatic system disorders) | 11 (21) | 13 (28)
Neutropenia (Blood and lymphatic system disorders) | 66 (173) | 76 (197)
Thrombocytopenia (Blood and lymphatic system disorders) | 22 (31) | 22 (45)
Hyperthyroidism (Endocrine disorders) | 23 (27) | 7 (8)
Hypothyroidism (Endocrine disorders) | 48 (58) | 20 (22)
Dry eye (Eye disorders) | 15 (15) | 9 (9)
Abdominal pain (Gastrointestinal disorders) | 16 (17) | 22 (24)
Abdominal pain upper (Gastrointestinal disorders) | 25 (28) | 29 (36)
Constipation (Gastrointestinal disorders) | 70 (95) | 61 (80)
Diarrhoea (Gastrointestinal disorders) | 146 (335) | 139 (278)
Dry mouth (Gastrointestinal disorders) | 13 (13) | 14 (15)
Dyspepsia (Gastrointestinal disorders) | 27 (29) | 27 (42)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12 (19) | 14 (17)
Haemorrhoids (Gastrointestinal disorders) | 16 (16) | 14 (15)
Nausea (Gastrointestinal disorders) | 145 (323) | 139 (287)
Stomatitis (Gastrointestinal disorders) | 51 (68) | 46 (56)
Vomiting (Gastrointestinal disorders) | 78 (115) | 53 (89)
Asthenia (General disorders) | 96 (193) | 87 (200)
Chills (General disorders) | 9 (9) | 14 (16)
Fatigue (General disorders) | 63 (107) | 38 (49)
Malaise (General disorders) | 12 (21) | 16 (21)
Mucosal inflammation (General disorders) | 32 (41) | 29 (42)
Oedema peripheral (General disorders) | 15 (22) | 16 (17)
Pain (General disorders) | 15 (20) | 17 (23)
Pyrexia (General disorders) | 44 (61) | 47 (73)
COVID-19 (Infections and infestations) | 8 (8) | 14 (14)
Conjunctivitis (Infections and infestations) | 14 (16) | 17 (17)
Nasopharyngitis (Infections and infestations) | 18 (21) | 15 (17)
Paronychia (Infections and infestations) | 14 (14) | 13 (16)
Upper respiratory tract infection (Infections and infestations) | 20 (24) | 21 (22)
Urinary tract infection (Infections and infestations) | 25 (35) | 24 (31)
Infusion related reaction (Injury, poisoning and procedural complications) | 39 (57) | 33 (42)
Procedural pain (Injury, poisoning and procedural complications) | 14 (14) | 18 (19)
Radiation skin injury (Injury, poisoning and procedural complications) | 52 (54) | 42 (43)
Wound complication (Injury, poisoning and procedural complications) | 13 (14) | 16 (16)
Alanine aminotransferase increased (Investigations) | 82 (138) | 65 (98)
Aspartate aminotransferase increased (Investigations) | 69 (105) | 51 (78)
Blood alkaline phosphatase increased (Investigations) | 11 (14) | 14 (16)
Blood lactate dehydrogenase increased (Investigations) | 12 (13) | 10 (10)
Ejection fraction decreased (Investigations) | 17 (17) | 19 (26)
Lymphocyte count decreased (Investigations) | 13 (21) | 12 (20)
Neutrophil count decreased (Investigations) | 33 (69) | 29 (47)
Platelet count decreased (Investigations) | 17 (23) | 13 (19)
Weight decreased (Investigations) | 26 (27) | 17 (17)
White blood cell count decreased (Investigations) | 13 (25) | 10 (16)
Decreased appetite (Metabolism and nutrition disorders) | 46 (62) | 35 (43)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 (16) | 4 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 12 (16) | 10 (12)
Hypomagnesaemia (Metabolism and nutrition disorders) | 12 (21) | 14 (22)
Arthralgia (Musculoskeletal and connective tissue disorders) | 59 (88) | 52 (79)
Back pain (Musculoskeletal and connective tissue disorders) | 23 (29) | 19 (21)
Bone pain (Musculoskeletal and connective tissue disorders) | 15 (16) | 19 (22)
Myalgia (Musculoskeletal and connective tissue disorders) | 45 (61) | 42 (66)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 (42) | 23 (31)
Dizziness (Nervous system disorders) | 23 (30) | 23 (30)
Dysgeusia (Nervous system disorders) | 33 (37) | 35 (40)
Headache (Nervous system disorders) | 53 (82) | 50 (69)
Hypoaesthesia (Nervous system disorders) | 14 (17) | 9 (11)
Neuropathy peripheral (Nervous system disorders) | 43 (50) | 45 (59)
Paraesthesia (Nervous system disorders) | 15 (16) | 20 (25)
Peripheral sensory neuropathy (Nervous system disorders) | 47 (56) | 40 (45)
Polyneuropathy (Nervous system disorders) | 14 (19) | 13 (15)
Anxiety (Psychiatric disorders) | 9 (9) | 14 (16)
Insomnia (Psychiatric disorders) | 39 (48) | 29 (36)
Dysuria (Renal and urinary disorders) | 19 (23) | 17 (21)
Breast pain (Reproductive system and breast disorders) | 11 (11) | 15 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 39 (50) | 48 (65)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (23) | 22 (33)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 32 (35) | 28 (38)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 13 (14)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 25 (29) | 14 (18)
Alopecia (Skin and subcutaneous tissue disorders) | 151 (158) | 146 (156)
Dermatitis (Skin and subcutaneous tissue disorders) | 22 (24) | 13 (14)
Dry skin (Skin and subcutaneous tissue disorders) | 23 (25) | 21 (22)
Erythema (Skin and subcutaneous tissue disorders) | 14 (20) | 17 (21)
Nail discolouration (Skin and subcutaneous tissue disorders) | 17 (17) | 25 (25)
Nail disorder (Skin and subcutaneous tissue disorders) | 18 (20) | 22 (23)
Onycholysis (Skin and subcutaneous tissue disorders) | 14 (16) | 6 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 36 (42) | 25 (35)
Rash (Skin and subcutaneous tissue disorders) | 63 (96) | 49 (62)
Hot flush (Vascular disorders) | 25 (29) | 25 (28)
Hypertension (Vascular disorders) | 14 (22) | 13 (21)

LIMITATIONS AND CAVEATS:
On February 5, 2021, the experimental treatment was discontinued and unblinded following the recommendation of the independent Data Monitoring Committee (iDMC) to stop treatment with atezolizumab/placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/79/NCT03726879/Prot_002.pdf
  • Statistical Analysis Plan (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT03726879/SAP_001.pdf